CLINICAL TRIAL: NCT01253200
Title: Clinical Evaluation of the Blazer® Open-Irrigated Radiofrequency Ablation Catheter for the Treatment of Type 1 Atrial Flutter
Brief Title: Clinical Evaluation of the Blazer® Open-Irrigated Catheter for Treatment of Type 1 Atrial Flutter
Acronym: BLOCk-CTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BLOCk-CTI
Record Dates: First submitted 2010-11-21; First posted 2010-12-03 (Estimated); Results first posted 2018-02-15 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-02

CONDITIONS: Atrial Flutter
Keywords: Type 1 Atrial Flutter; Typical Atrial Flutter; Arrhythmias, Cardiac; Heart Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Atrial Flutter; Arrhythmias, Cardiac; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Masking Description: Subject was not told by investigator if device used was Investigational or Control. The subject could ask the investigator at end of study at 3 months if they wanted to know which device was used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Blazer® Open-Irrigated Ablation Catheter (Experimental): Patients treated with the Blazer® Open-Irrigated Ablation Catheter
  Interventions: Device: Blazer® Open-Irrigated Ablation Catheter
- Control Catheter (Active Comparator): Patients treated with an open-irrigated radiofrequency ablation catheter that has received FDA market approval for the treatment of type 1 atrial flutter( Biosense Webster ThermoCool® ablation catheters (NaviStar™, EZ Steer, or SF) or St. Jude Medical ablation catheters (Therapy™ Cool Path™ or Safire BLU™),
  Interventions: Device: Control Catheter

INTERVENTIONS:
Device: Blazer® Open-Irrigated Ablation Catheter — Blazer® Open-Irrigated Ablation Catheter
  Arms: Blazer® Open-Irrigated Ablation Catheter
Device: Control Catheter — Open-irrigated radiofrequency ablation catheters that have received FDA market approval for the treatment of type 1 atrial flutter
  Other Names: ThermoCool, NaviStar, EZ Steer, SF, Cool Path, Safire BLU
  Arms: Control Catheter

SUMMARY:
The purpose of the BLOCk-CTI study is to evaluate the safety and effectiveness of the Blazer® Open-Irrigated Ablation Catheter for the treatment of sustained or recurrent type 1 atrial flutter. This study will compare outcomes in patients treated with the Blazer® Open-Irrigated Ablation Catheter to outcomes in patients treated with open-irrigated radiofrequency ablation catheters that have received FDA market approval for the treatment of type 1 atrial flutter.

DETAILED DESCRIPTION:
The BLOCk-CTI study is a prospective, multicenter, single blind, 1:1 randomized study. The study is designed to demonstrate that the safety and effectiveness of the Blazer® Open-Irrigated Ablation Catheter are non-inferior to the safety and effectiveness of the control catheters. In this study, the control catheters are open-irrigated radiofrequency ablation catheters that have received FDA market approval for the treatment of type 1 atrial flutter. (Biosense Webster ThermoCool® ablation catheters (NaviStar™, EZ Steer, or SF) or St. Jude Medical ablation catheters (Therapy™ Cool Path™ or Safire BLU™).

ELIGIBILITY:
Inclusion Criteria:

* At least 1 documented episode of type 1 atrial flutter in the 180 days (6 months) preceding enrollment documented by 12-lead ECG, Holter monitor, rhythm strip, or transtelephonic monitor
* Patients are clinically indicated for catheter ablation
* Patients receiving oral anti-arrhythmic drug therapy (class I or class III) for a tachyarrhythmia other than type 1 atrial flutter must be controlled on the anti-arrhythmic drug for a minimum of 30 days prior to enrollment. If type 1 atrial flutter was documented prior to the development of other tachyarrhythmias, this 30-day period is not required.
* Age 18 or above, or of legal age to give informed consent specific to state and national law
* Patients are competent and willing to provide written informed consent to participate in the study and agree to comply with follow-up visits and evaluation

Exclusion Criteria:

* Any prior right atrial cavo-tricuspid isthmus ablation or any cardiac ablation for non-atrial flutter arrhythmias within 90 days prior to enrollment
* Cardiac surgery within 90 days prior to enrollment
* Myocardial infarction within 60 days prior to enrollment
* Current unstable angina
* Patients who cannot have anti-arrhythmic drugs (class I and class III) prescribed for the treatment of type 1 atrial flutter stopped on the day of the procedure
* Patients regularly prescribed amiodarone within the 120 days (4 months) prior to enrollment
* Documented atrial or ventricular tumors, clots, thrombus, or have a known clotting disorder within 90 days prior to enrollment
* Implantation of permanent leads of an implantable device in or through the right atrium within 90 days prior to enrollment
* Direct remedial cause of atrial flutter (e.g. thyroid disease, pericarditis, pulmonary embolic disease)
* Atypical or scar-based flutter
* Patients with New York Heart Association Class III at the time of enrollment or New York Heart Association Class IV heart failure within 90 days prior to enrollment
* Patients with an ejection fraction less than 30% within 90 days prior to enrollment
* Clinically significant structural heart disease (including tricuspid valve regurgitation, tricuspid valve stenosis, tricuspid valve replacement, Ebstein's anomaly, or other congenital heart disease) that would preclude catheter introduction and placement, as determined by the Investigator
* Any cerebral ischemic event (including transient ischemic attacks) within 180 days prior to enrollment
* Contraindication to anticoagulation therapy based upon published guidelines
* Creatinine greater than 2.5 mg/dl or creatinine clearance less than 30 mL/min within 90 days prior to enrollment
* Any other significant uncontrolled or unstable medical condition (e.g. sepsis, acute metabolic illness)
* Enrolled in any concurrent study without BSC written approval
* Women who are pregnant or plan to become pregnant within the course of their participation in the investigation
* Life expectancy less than or equal to 2 years (730 days) per physician opinion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2011-01; Primary Completion 2013-09 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tom McElderry, MD, Principal Investigator — University of Alabama at Birmingham
Locations (26):
- United States (26):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - St. Jude Medical Center, Fullerton, California
  - Regional Cardiology Associates, Sacramento, California
  - Colorado Springs Cardiologist, P.C., Colorado Springs, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - West Coast Arrhythmia Center, Hudson, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Georgia Health Sciences University, Augusta, Georgia
  - University of Kansas Hospital, Kansas City, Kansas
  - Central Baptist Hospital, Lexington, Kentucky
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Caritas St. Elizabeth's Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Strong Memorial Hospital of the University of Rochester, Rochester, New York
  - Moses H. Cone Memorial Hospital, Greensboro, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - ProMedica Toledo Hospital, Toledo, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Cardiac Arrhythmia Research, Austin, Texas
  - Hall Garcia Cardiology, Houston, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Swedish Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from referring physicians for ablation for type 1 atrial flutter
Pre-assignment Details: Subjects were excluded if there were no documented episodes of atrial flutter or inclusion criteria were not met. Roll-in subjects were not randomized.
Groups:
- Randomized Blazer® Open-Irrigated Ablation Catheter: Randomized Patients treated with the Blazer® Open-Irrigated Ablation Catheter
  Blazer® Open-Irrigated Ablation Catheter: Blazer® Open-Irrigated Ablation Catheter
- Randomized Control Catheter: Randomized patients treated with an open-irrigated radiofrequency ablation catheter that has received FDA market approval for the treatment of type 1 atrial flutter
  Control Catheter: Open-irrigated radiofrequency ablation catheters that have received FDA market approval for the treatment of type 1 atrial flutter
- Roll-in Blazer Open Irrigated Subjects: The use of the Blazer-Open Irrigated Catheter was required after the second study suspension. Previously enrolled subjects prior to suspension were also classified as Roll-in subjects; not counted in endpoint analysis.
- Roll-in Control Catheter: The use of the Control Catheter was optional after the second study suspension in a Roll-in subject. Previously enrolled subjects prior to suspension were also classified as Roll-in subjects; not counted in endpoint analysis.
- Not Randomized to Any Treatment Group Subjects: Five subjects were not Randomized to any treatment group and were not Roll-in subjects.
Period: Overall Study
Arm/Group | Randomized Blazer® Open-Irrigated Ablation Catheter | Randomized Control Catheter | Roll-in Blazer Open Irrigated Subjects | Roll-in Control Catheter | Not Randomized to Any Treatment Group Subjects
Started | 125 | 125 | 30 | 17 | 5
Procedure | 109 | 111 | 28 | 12 | 0
10 Day Follow-up | 106 | 111 | 28 | 12 | 0
3 Month Follow-up | 104 | 106 | 28 | 12 | 0
Completed | 104 | 106 | 28 | 12 | 0
Not Completed | 21 | 19 | 2 | 5 | 5
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 4 | 0 | 0 | 5
Not completed — intents | 10 | 10 | 1 | 3 | 0
Not completed — Attempts | 6 | 4 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Randomized Blazer® Open-Irrigated Ablation Catheter: Patients randomized to treatment with the Blazer® Open-Irrigated Ablation Catheter
- Randomized Control Catheter: Patients randomized to treatment with an open-irrigated radiofrequency ablation catheter that has received FDA market approval for the treatment of type 1 atrial flutter
  Control Catheter: Open-irrigated radiofrequency ablation catheters that have received FDA market approval for the treatment of type 1 atrial flutter
- Roll-In Blazer® Open-Irrigated Ablation Catheter: The use of the Blazer-Open Irrigated Catheter was required after the second study suspension. Previously enrolled subjects prior to suspension were also classified as Roll-in subjects; not counted in endpoint analysis.
- Not Randomized to Any Treatment Group: Subjects not Randomized to any treatment group and were not Roll-in subjects
- Total: Total of all reporting groups
Arm/Group | Randomized Blazer® Open-Irrigated Ablation Catheter | Randomized Control Catheter | Roll-In Blazer® Open-Irrigated Ablation Catheter | Roll-In Control Catheter | Not Randomized to Any Treatment Group | Total
Number analyzed (Participants) | 125 | 125 | 30 | 17 | 5 | 302
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (11) | 66 (10) | 69 (10) | 66 (9) | 72 (11) | 65.73 (10.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 29 | 4 | 4 | 2 | 62
  Male | 102 | 96 | 26 | 13 | 3 | 240
Region of Enrollment [Number; unit: participants]
  United States | 125 | 125 | 30 | 17 | 5 | 302

OUTCOME MEASURES:

1. Primary Outcome: Procedure-related Complication-free Rate
Description: A procedure-related complication is defined as an adverse event that results in death, a life-threatening complication, or a persistent or significant disability/incapacity or required intervention to prevent a permanent impairment of a body function or damage to a body structure. All adverse events related to the investigational or control devices or ablation procedure will be considered procedure-related events.
Time Frame: 7 days post-procedure
Population: The primary outcome analysis is for a further subset of Randomized subjects only who underwent RF ablation; 220 subjects out of the total 302 subjects. All is consistent with the approved statistical analysis plan and information publicly available in the FDA Summary of Safety and Effectiveness Data (SSED) and BSC labeling, the Directions for Use.
Measure: Number; unit: percentage of subjects
Groups:
- Control Catheter: Patients treated with an open-irrigated radiofrequency ablation catheter that has received FDA market approval for the treatment of type 1 atrial flutter
  Control Catheter: Open-irrigated radiofrequency ablation catheters that have received FDA market approval for the treatment of type 1 atrial flutter
Arm/Group | Blazer® Open-Irrigated Ablation Catheter | Control Catheter
Number analyzed (Participants) | 109 | 111
percentage of subjects | 92.7 | 98.2
Statistical Analysis 1: Comparison: Blazer® Open-Irrigated Ablation Catheter vs Control Catheter; Note that analysis of the primary outcome was conducted for Randomized subjects only as prespecified in the study protocol. This is consistent analysis publicly available in the Summary of Safety and Effectiveness Data (SSED); Test type: Non-Inferiority or Equivalence — The Primary Safety Endpoint was evaluated using a one-sided, non-inferiority test for two binomial proportions at an alpha-level of 0.05. A 95% confidence interval based upon a score test of the difference of proportion of subjects in the Investigational and Control Groups free from a procedure-related complication seven days post-procedure was constructed. The upper bound of the confidence interval was compared to 10%; Risk Difference (RD) = 4.6, 95% CI 1-sided [upper limit 9.78]

2. Primary Outcome: Acute Success Rate
Description: Acute success is defined as demonstration of bidirectional cavo-tricuspid isthmus block (ie, lack of electrophysiological conduction through the isthmus) 30 minutes after the last radiofrequency application in the cavo-tricuspid isthmus with the investigational or control catheter only.
Time Frame: 30 minutes after the last radiofrequency application in the cavo-tricuspid isthmus
Population: as for outcome 1
Measure: Number; unit: percentage of success
Arm/Group | Blazer® Open-Irrigated Ablation Catheter | Control Catheter
Number analyzed (Participants) | 109 | 111
percentage of success | 87.2 | 89.2

3. Secondary Outcome: Chronic Success Rate: All Treated Patients
Description: Chronic success is defined as freedom from recurrence of type 1 atrial flutter at 3-months post-procedure for all treated patients.
Time Frame: 3 months post-procedure
Population: The secondary outcome analysis is for a subset of Randomized subjects only who underwent RF ablation; 220 subjects out of the total 302 subjects. All is consistent with the approved statistical analysis plan and information publicly available in the FDA Summary of Safety and Effectiveness Data (SSED) and BSC labeling, the Directions for Use.
Measure: Number; unit: percentage of subjects
Arm/Group | Blazer® Open-Irrigated Ablation Catheter | Control Catheter
Number analyzed (Participants) | 109 | 111
percentage of subjects | 74.3 | 80.2

4. Secondary Outcome: Chronic Success Rate: Acute Success Patients
Description: Chronic success is defined as demonstration of acute success and freedom from recurrence of type 1 atrial flutter at 3-months post-procedure. Only randomized patients with acute procedural success will be included in this endpoint.
Time Frame: 3-months post-procedure
Population: The secondary outcome analysis is for a further subset of Randomized subjects only who underwent RF ablation and classified as acute success; 194 of the total 302 subjects. All consistent with approved statistical analysis plan and information publicly available in the FDA SSED and BSC the Directions for Use.
Measure: Number; unit: percentage of chronic success
Arm/Group | Blazer® Open-Irrigated Ablation Catheter | Control Catheter
Number analyzed (Participants) | 95 | 99
percentage of chronic success | 85.3 | 89.9

ADVERSE EVENTS:
Time Frame: Within 3 months of the index RF ablation procedure
Description: Only subjects at risk for adverse events, (Randomized and Roll-in for the Blazer Open-irrigated catheter and the Control Catheters) are included in the calculation of the adverse event rate. The calculation of the adverse event rate does NOT include the five Non-randomized subjects who were NOT treated with either the Blazer Open-irrigated catheter or the Control Catheter.
Groups:
- Randomized Blazer® Open-Irrigated Ablation Catheter: Randomized patients treated with the Blazer® Open-Irrigated Ablation Catheter (procedure patients)
  Blazer® Open-Irrigated Ablation Catheter: Blazer® Open-Irrigated Ablation Catheter
  Note that only subjects at risk for an adverse event (treated subjects) are included in the calculation of the adverse event rates
- Randomized Control Catheter: Randomized patients treated with an open-irrigated radiofrequency ablation catheter that has received FDA market approval for the treatment of type 1 atrial flutter (procedure patients)
  Control Catheter: Open-irrigated radiofrequency ablation catheters that have received FDA market approval for the treatment of type 1 atrial flutter
  Note that only subjects at risk for an adverse event (treated subjects) are included in the calculation of the adverse event rates
- Roll-in Blazer® Open-Irrigated Ablation Catheter: Roll-in patients treated with the Blazer® Open-Irrigated Ablation Catheter (procedure patients)
  Blazer® Open-Irrigated Ablation Catheter: Blazer® Open-Irrigated Ablation Catheter
  Note that only subjects at risk for an adverse event (treated subjects) are included in the calculation of the adverse event rates
- Roll-in Control Catheter: Roll-in patients treated with an open-irrigated radiofrequency ablation catheter that has received FDA market approval for the treatment of type 1 atrial flutter (procedure patients)
  Control Catheter: Open-irrigated radiofrequency ablation catheters that have received FDA market approval for the treatment of type 1 atrial flutter
  Note that only subjects at risk for an adverse event (treated subjects) are included in the calculation of the adverse event rates
- Non-Randomized to Any Treatment Group: Five subjects were not randomized to any treatment group and were not Roll-in subjects. Therefore, these five subjects were not treated with the Blazer Open-irrigated catheter or a Control catheter.
  Note that only subjects at risk for an adverse event (treated subjects) are included in the calculation of the adverse event rates
Arm/Group | Randomized Blazer® Open-Irrigated Ablation Catheter | Randomized Control Catheter | Roll-in Blazer® Open-Irrigated Ablation Catheter | Roll-in Control Catheter | Non-Randomized to Any Treatment Group
All-Cause Mortality (participants affected / at risk) | 1/125 | 0/125 | 0/30 | 0/17 | 0/5
Serious Adverse Events (participants affected / at risk) | 7/109 | 2/111 | 5/28 | 2/12 | 0/5
Other Adverse Events (participants affected / at risk) | 50/109 | 61/111 | 16/28 | 7/12 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Blazer® Open-Irrigated Ablation Catheter (N=109) | Randomized Control Catheter (N=111) | Roll-in Blazer® Open-Irrigated Ablation Catheter (N=28) | Roll-in Control Catheter (N=12) | Non-Randomized to Any Treatment Group (N=5)
Cardiovascular Accident (CVA) Resulting in Death (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Cardiovascular Accident (CVA) Resulting in Death
Hypotension (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Hypotension
Congestive Heart Failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Congestive Heart Failure
Vasovagal Reaction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — syncope
Junctional Rhythm (Cardiac disorders) | 1 (1) | 0 | 0 (0) | 0 (0) | 0 (0) — Junctional Rhythm Requiring Pacemaker Implantation
Pseudoaneurysm with Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Pseudoaneurysm with Hematoma
Pseudoaneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Pseudoaneurysm
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Urinary Tract Infection
3rd Degree Heart Block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — AF
Chest pain iscemic (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial perforation with tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nonsustained ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — NSVT
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Blazer® Open-Irrigated Ablation Catheter (N=109) | Randomized Control Catheter (N=111) | Roll-in Blazer® Open-Irrigated Ablation Catheter (N=28) | Roll-in Control Catheter (N=12) | Non-Randomized to Any Treatment Group (N=5)
Ablation related Events (Cardiac disorders) | 6 (7) | 12 (13) | 3 (3) | 2 (2) | 0 (0) — events related to ablation procedure
Cardiovascular related (Cardiac disorders) | 41 (56) | 52 (97) | 14 (18) | 5 (5) | 0 (0) — arrhythmias, chest pain, CVA, symptoms
Non-cardiovascular (General disorders) | 11 (12) | 11 (16) | 4 (4) | 1 (1) | 0 (0) — Non-cardiovascular

LIMITATIONS AND CAVEATS:
Two interim study suspensions occurred during enrollment that did not impact the integrity of the data and subsequent analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No